CLINICAL TRIAL: NCT06723353
Title: Effects of Visceral Manipulation Combined with Kinesio Taping on Diastasis Recti, Pain Intensity, Stress Incontinence, Pelvic Floor Strength, and Overall Wellness in Postpartum Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Health and Research-Insights (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LUC/CPGS/PHDE/PTR/20240329/001
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Diastasis Recti; Diastasis Recti Abdominis (DRA)
Keywords: Diastasis Recti Abdominis (DRA); Postpartum Recovery; Visceral Manipulation (VM); Kinesio Taping (KT); Core Strengthening Exercises; Pelvic Floor Dysfunction; Inter-Recti Distance (IRD); Urinary Incontinence; Pain Management; Physical Therapy for Postpartum Women
MeSH Terms: conditions — Urinary Incontinence; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Visceral Manipulation (Experimental): Participants in this arm will receive Visceral Manipulation (VM) therapy administered by a trained physical therapist. VM is a gentle manual therapy aimed at releasing restrictions within the visceral system to improve the mobility and function of the internal organs. The therapy sessions will focus on enhancing abdominal organ mobility and will be performed in a clinical setting. This treatment will be administered over a six-week period with sessions occurring once per week.
  Interventions: Other: Visceral Manipulation Therapy
- Kinesio Taping (Experimental): This arm involves the application of Kinesio Tape (KT) to the abdominal area to support and stabilize the muscles affected by Diastasis Recti Abdominis. The KT will be applied in a crisscross manner to potentially facilitate muscle function and reduce the Inter-Recti Distance (IRD). Participants will receive taping once a week for six weeks, and the tape will be maintained throughout the week to ensure continuous support.
  Interventions: Other: Abdominal Kinesio Taping
- Combined Visceral Manipulation and Kinesio Taping (Experimental): Participants in this arm will receive a combination of Visceral Manipulation and Kinesio Taping. The combination is intended to maximize the therapeutic effects by enhancing organ function with VM and providing muscular support with KT. The treatments will be administered concurrently during the same six-week period, with weekly sessions for both therapies.
  Interventions: Other: Combined Visceral Manipulation and Kinesio Taping
- Core Strengthening Exercises (Active Comparator): This arm involves participants engaging in core strengthening exercises specifically designed for postpartum rehabilitation. The exercises aim to strengthen the transverse abdominis, multifidus, and pelvic floor muscles, which support the abdominal organs and improve core stability. Participants will perform these exercises under the supervision of a physical therapist three times a week for six weeks to ensure proper technique and progression.
  Interventions: Other: Postpartum Core Strengthening Program

INTERVENTIONS:
Other: Visceral Manipulation Therapy — Visceral Manipulation (VM) is a manual therapy consisting of gentle, specifically placed manipulations that encourage normal mobility, tone, and inherent tissue motion of the viscera and their connective tissues. These manipulations can potentially improve the structural integrity of the abdominal cavity and enhance the physiological functioning of the organs. VM will be administered by certified therapists trained in this specialized technique, focusing on reducing the Inter-Recti Distance (IRD) and associated symptoms of DRA.
  Arms: Visceral Manipulation
Other: Abdominal Kinesio Taping — Kinesio Taping (KT) involves the application of a thin, stretchable tape over and around muscles to enhance function, reduce inflammation, and support muscles in movement on a 24hr/day basis. It is non-restrictive, allowing for full range of motion. In this study, KT will be applied in a crisscross pattern across the abdomen to support the abdominal muscles affected by DRA, potentially aiding in muscle function and reducing pain and discomfort.
  Arms: Kinesio Taping
Other: Combined Visceral Manipulation and Kinesio Taping — This intervention combines Visceral Manipulation and Kinesio Taping to leverage the benefits of both modalities. The combination aims to enhance the functional and structural support of the abdominal region by improving organ function through VM and providing muscular support through KT. This dual approach is hypothesized to offer a synergistic benefit, potentially providing a more effective treatment for reducing IRD and improving overall abdominal function.
  Arms: Combined Visceral Manipulation and Kinesio Taping
Other: Postpartum Core Strengthening Program — The Core Strengthening Program is designed to strengthen the deep core muscles, including the transverse abdominis, multifidus, and the pelvic floor muscles. Exercises will be tailored to accommodate postpartum women and will be progressively adjusted to match improvements in strength and endurance. The program includes supervised training sessions focusing on enhancing core stability, which is crucial for postpartum recovery and long-term spinal and pelvic health.
  Arms: Core Strengthening Exercises

SUMMARY:
This clinical trial aims to evaluate the effectiveness of different therapies for treating Diastasis Recti Abdominis (DRA) in postpartum women. DRA, commonly experienced after childbirth, involves the separation of abdominal muscles, which can lead to discomfort and decreased core stability. The main questions this study seeks to answer are:

How effective are Visceral Manipulation (VM), Kinesio Taping (KT), and core strengthening exercises in reducing the gap between abdominal muscles (Inter-Recti Distance or IRD)? Do these treatments improve pain levels, pelvic floor muscle strength, and urinary incontinence? This study will compare the effects of VM, KT, a combination of both, and core strengthening exercises to determine which therapy-or combination of therapies-most effectively treats DRA.

Participants will:

Be randomly assigned to one of four treatment groups: VM, KT, VM combined with KT, or core strengthening exercises.

Undergo their designated treatments for a period of 6 weeks. Visit the clinic for assessments at the start, mid-point, and end of the treatment period.

Complete surveys and undergo physical tests to measure changes in IRD, pain levels, pelvic floor strength, and urinary function.

This research will provide valuable insights into the most effective treatments for DRA, aiming to enhance the well-being and recovery of postpartum women.

DETAILED DESCRIPTION:
Overview

This clinical trial is designed to investigate the efficacy of various interventions in treating Diastasis Recti Abdominis (DRA) among postpartum women. DRA is a condition characterized by the separation of the left and right sides of the rectus abdominis muscle, commonly occurring during and after pregnancy. This separation can lead to functional impairments such as lower back pain, pelvic floor dysfunctions, and a decrease in core stability, which significantly affects a woman's quality of life.

Purpose

The study aims to assess and compare the effectiveness of four different treatment modalities: Visceral Manipulation (VM), Kinesio Taping (KT), a combination of both VM and KT, and core strengthening exercises. The primary goal is to determine which treatment(s) most effectively reduce the inter-recti distance (IRD), thus alleviating the physical and functional symptoms associated with DRA. Secondary objectives include evaluating the impact of these treatments on associated pain levels, pelvic floor muscle strength, and urinary incontinence, which are common concerns among affected postpartum women.

Study Design

This randomized controlled trial will enroll participants from four major maternity hospitals across Karachi, Pakistan, ensuring a diverse participant pool. Upon meeting inclusion criteria, participants will be randomly assigned to one of the four intervention groups. Each group will receive a specific treatment protocol for six weeks, with assessments scheduled at baseline, the three-week midpoint, and upon completion at six weeks.

Group A: Participants will receive Kinesio Taping applied with approximately 70% tension in a crisscross pattern over the rectus abdominis muscle.

Group B: Participants will undergo Visceral Manipulation, focusing on enhancing the mobility and function of abdominal and pelvic organs.

Group C: This group will receive both VM and KT as combined therapies to maximize the therapeutic benefits.

Group D: Participants in this group will perform targeted core strengthening exercises designed to enhance muscle function and support abdominal healing.

Methodology

Treatment efficacy will be evaluated through a series of quantitative and qualitative measurements:

Inter-Recti Distance (IRD): Measured using the finger-width palpation method, this metric will directly assess the physical gap between the rectus abdominis muscles.

Pain Level: Assessed using the Visual Analogue Scale (VAS), allowing participants to report the intensity of their pain.

Pelvic Floor Muscle Strength: Evaluated using pressure biofeedback units, providing objective data on muscle functionality.

Urinary Incontinence: Measured via the Urinary Distress Inventory-6 (UDI-6), which quantifies symptoms of urinary incontinence.

Data Analysis

Data will be processed and analyzed using the Statistical Package for the Social Sciences (SPSS), version 21.0. Analysis of Covariance (ANCOVA) will be used to compare treatment effects across the groups, adjusting for potential confounders like age and BMI. Repeated measures ANOVA will be employed to evaluate changes within each group over time.

Ethical Considerations

The study has been reviewed and approved by an Institutional Review Board, ensuring that all procedures adhere to ethical guidelines. Participants will provide informed consent before participating, with a guarantee of confidentiality and the right to withdraw from the study at any time without penalty.

Significance

By rigorously evaluating these interventions, the study aims to provide clear, evidence-based guidance on the most effective treatment strategies for managing DRA in postpartum women. This research is crucial not only for enhancing individual patient care but also for informing clinical practices and potentially influencing public health policies related to maternal health and recovery.

ELIGIBILITY:
Inclusion Criteria:

Post-partum female will be included on the basis of:

* DRA: Finger width palpation shows >2.5 cm
* Postpartum females bearing at least 1 child
* Age between 35 to 45 years old
* Post-partum females who had gone through normal vaginal delivery, vacuum delivery, forceps delivery, and lower section caesarian section (at least 1 month after)

Exclusion Criteria:

Postpartum female will be excluded if she has:

* Any other abdominal surgery
* Sensitivity with taping (specific for those will have KT)
* Diagnosed with abdominal hernia
* Open abdominal wound

Ages: 35 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Reduction in Inter-Recti Distance (IRD) | Baseline, at the end of 3 weeks (mid-intervention), and at the end of 6 weeks (post-intervention)
  This measure assesses the effectiveness of the interventions in reducing the Inter-Recti Distance (IRD) between the rectus abdominis muscles. The IRD will be measured using the finger-width palpation method, which involves placing fingers horizontally across the midline of the participant's abdomen at, above, and below the umbilicus. This method provides a direct and tangible measure of the gap between the rectus abdominis muscles, which is a primary physical manifestation of Diastasis Recti Abdominis (DRA).

SECONDARY OUTCOMES:
Improvement in Pelvic Floor Muscle Strength | Baseline, at the end of 3 weeks (mid-intervention), and at the end of 6 weeks (post-intervention)
  This secondary outcome measure evaluates the effectiveness of the interventions in enhancing the strength and functionality of pelvic floor muscles. Strength will be quantified using pressure biofeedback units, which provide precise measurements of muscle contraction and relaxation. This assessment is crucial for understanding the broader impact of the interventions on postpartum pelvic health, which is often compromised in cases of DRA.

CONTACTS AND LOCATIONS:
Locations (1):
- Jinnah Postgraduate Medical Center, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) from this study will not be shared publicly due to concerns over privacy and confidentiality, particularly given the sensitive nature of the health data involved. This decision aligns with the participant consent terms, which specified that data would be used solely for this research. Ethical considerations also dictate maintaining control over the data to ensure integrity and prevent potential misuse. Additionally, logistical limitations regarding the infrastructure necessary for secure data management preclude public sharing. This approach ensures compliance with ethical standards and protects participant trust and data security.